CLINICAL TRIAL: NCT01805778
Title: Novel Approaches to the Prediction, Diagnosis and Treatment of Cardiac Late Effects in Survivors of Childhood Cancer: A Multi-centre Observational Study
Brief Title: Preventing Cardiac Sequelae in Pediatric Cancer Survivors
Acronym: PCS2
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Institute for Cancer Research (Other); Pediatric Oncology Group of Ontario (Other); C17 Council (Other); Ottawa Heart Institute Research Corporation (Other); Montreal Heart Institute (Other); McMaster Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); London Health Sciences Centre (Other); Children's Hospital of Orange County (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Principal Investigator, Paul Nathan, Director- Aftercare Program, Staff Oncologist, The Hospital for Sick Children
Other Study IDs: 1000032746
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Anthracycline-induced Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will retain plasma for biomarker and genomic analysis. The study will also retain saliva for those patient who are unable or unwilling to provide a blood specimen for genomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute Cohort: Patients newly diagnosed with cancer who will be receiving anthracycline chemotherapy
- Survivor Cohort: Survivors of childhood cancer who are at least 3 years or more from their last dose of anthracycline therapy.

SUMMARY:
Cancer therapy can place childhood cancer survivors at increased risk for heart disease which can lead to significant illness or early death. Interventions that occur late in the evolution of treatment-related heart disease are usually ineffective at preventing its progression to death or heart transplant. Our team will work in several research cores to test new imaging and biomarker methods that will lead to earlier detection of heart disease before clinical symptoms develop or it become apparent on standard imaging tests. We will evaluate the importance of genetic differences between individuals in determining who is at greatest risk of developing heart disease as a result of exposure to cardiotoxic agents. We will combine this genetic information with the novel imaging and biomarker methods to predict which children are at particular risk. These vulnerable children can then be targeted by modifying their cancer therapy to reduce their exposure to cardiac toxins, or introducing medications that protect the heart from chemotherapy damage. This team brings together the expertise of clinicians and scientists in pediatric oncology, pediatric and adult cardiology, radiation oncology, genetics, and biostatistics. This is a cross-Canada initiative that will leverage the latest knowledge about cardiac toxicity and create a resource for ongoing research into this important cause of morbidity and mortality in childhood cancer survivors.

DETAILED DESCRIPTION:
This is a multi-centre observational cohort study that will be conducted at The Hospital for Sick Children (Toronto), Princess Margaret Hospital (Toronto), McMaster Children's Hospital (Hamilton), London Health Sciences Centre (London), The Children's Hospital of Eastern Ontario (Ottawa) and The Children's Hospital of Orange County (Orange County, California).

The study will address the current limitations in prediction and early diagnosis of anthracycline-induced heart disease. This will be accomplished by the following 3 collaborative cores:

Core 1 (Genomics) will focus on determining which children are most susceptible to treatment-related cardiac toxicity by assessing genes in pathways related to anthracycline absorption, distribution, metabolism, and excretion, as well identifying genes in pathways known to be important in the cardiac response to injury.

Core 2 (Biomarkers) will explore whether existing and novel biomarkers allow for more accurate diagnosis of acute and late treatment-related cardiac toxicity. The core will use a human stem cell platform for discovery of novel biomarkers of anthracycline cardiac damage that will be evaluated in our clinical cohort.

Core 3 (Cardiac imaging) will focus on the evaluation of new echocardiographic and CMR techniques aimed at early identification of cardiac damage after anthracycline exposure.

It will investigate whether changes in cardiac function immediately after anthracycline administration predict which patients will develop progressive cardiac disease over time, and it will explore disease progression through the longitudinal evaluation of innovative echocardiographic parameters of remodeling and dysfunction in CCS exposed to anthracyclines.

ELIGIBILITY:
ACUTE COHORT:

Inclusion Criteria:

* Aged <18 years at time of cancer diagnosis
* Diagnosed with a new malignancy (patients with a history of a prior malignancy wlil be eligible if they have not received any anthracycline chemotherapy or chest radiation)
* Cancer treatment plan will require therapy with at least one dose of any anthracycline
* Planned to have all pre-anthracycline echocardiograms (ECHO) at the recruiting site
* Normal cardiac functioning prior to initiation of anthracycline therapy (LV EF > 55%)
* Patients who are uncooperative during the ECHO without sedation or anesthesia will be included in the study. However, these patients will only undergo clinically indicated echocardiograms, with no echocardiograms added for purely research purposes
* Provision of signed informed consent by the patient and/or patient's legal guardian

Exclusion Criteria:

* Patients who were previously treated with anthracycline chemotherapy or radiation to the chest.
* Significant congenital heart defects, including patients with any other congenital cardiac abnormality, except those with a patent foramen ovale or a small ASD. Patients with familial cardiomyopathies (hypertrophic, dilated and restrictive) will be excluded.

SURVIVOR COHORT:

Inclusion Criteria:

* Aged < 18 years at time of cancer diagnosis
* Previously diagnosed with cancer and currently in remission
* Patients whose prior treatment plan included therapy with at least one dose of any anthracycline
* Patients who completed their final dose of anthracycline at least 3 years ago
* Routinely followed at the recruiting site approximately ever 12 months

Exclusion Criteria

* Prior allogeneic stem cell transplant
* Significant congenital heart defects, including patients with any other congenital cardiac abnormality, except those with a patent foramen ovale or a small ASD. Patients with familial cardiomyopathies (hypertrophic, dilated and restrictive) will be excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from pediatric oncology centres across Ontario, Canada (SickKids in Toronto, McMaster Children's Hospital in Hamilton, Children's Hospital of Eastern Ontario in Ottawa, and London Health Sciences Centre in London) as well as Princess Margaret Cancer Centre (Toronto) and Children's Hospital of Orange County (California, U.S.).
Sampling Method: Non-Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Cardiac Remodeling | one year after last dose of anthracycline therapy in Acute Cohort; anytime during 2 year follow up in Survivor Cohort
  The presence of one or more of the following:
  1. Cardiac Remodeling defined as Left Ventricular Posterior Wall Thickness (LVPWT) or Thickness to Dimension Ratio (TDR) z-score <-2.0 or a reduction in LVPWT or TDR z-score by at least 1 standard deviation compared to baseline; or
  2. Reduced left ventricular ejection fraction (LV EF) (<55%); or
  3. Symptomatic heart failure graded using New York Heart Association (NYHA) classification (or Ross heart failure class at least 2 in infants less than 2 years old)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Nathan, M.D., Principal Investigator — The Hospital for Sick Children; Mark Greenberg, M.D., Principal Investigator — The Hospital for Sick Children; Seema Mital, M.D., Principal Investigator — The Hospital for Sick Children; Luc Mertens, M.D., Principal Investigator — The Hospital for Sick Children; Paul Kantor, M.D., Principal Investigator — University of Alberta/Stollery Children's Hospital; Peter Liu, M.D., Principal Investigator — Ottawa Heart Institute
Locations (6):
- Children's Hospital of Orange County, Orange, California, United States
- Canada (5):
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - SickKids, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Chaix MA, Parmar N, Kinnear C, Lafreniere-Roula M, Akinrinade O, Yao R, Miron A, Lam E, Meng G, Christie A, Manickaraj AK, Marjerrison S, Dillenburg R, Bassal M, Lougheed J, Zelcer S, Rosenberg H, Hodgson D, Sender L, Kantor P, Manlhiot C, Ellis J, Mertens L, Nathan PC, Mital S. Machine Learning Identifies Clinical and Genetic Factors Associated With Anthracycline Cardiotoxicity in Pediatric Cancer Survivors. JACC CardioOncol. 2020 Dec 15;2(5):690-706. doi: 10.1016/j.jaccao.2020.11.004. eCollection 2020 Dec. PMID 34396283
- [Derived] Skitch A, Mital S, Mertens L, Liu P, Kantor P, Grosse-Wortmann L, Manlhiot C, Greenberg M, Nathan PC. Novel approaches to the prediction, diagnosis and treatment of cardiac late effects in survivors of childhood cancer: a multi-centre observational study. BMC Cancer. 2017 Aug 3;17(1):519. doi: 10.1186/s12885-017-3505-0. PMID 28774277